CLINICAL TRIAL: NCT00632229
Title: Double Blinded, Placebo-Controlled Trial of Paliperidone Addition in SRI-Resistant Obsessive-Compulsive Disorder
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University of South Florida (Other)
Collaborators: Indiana University (Other); Ortho-McNeil Janssen Scientific Affairs, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: USF 08-0100
Record Dates: First submitted 2008-02-29; First posted 2008-03-10 (Estimated); Results first posted 2014-02-06 (Estimated); Last update posted 2014-02-06 (Estimated); Status verified 2013-10

CONDITIONS: Obsessive-Compulsive Disorder
Keywords: Obsessive-Compulsive Disorder; Adults; Medication; Treatment
MeSH Terms: conditions — Obsessive-Compulsive Disorder | interventions — Paliperidone Palmitate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Paliperidone (Experimental): Recieves study medication called paliperidone
  Interventions: Drug: Paliperidone
- Pill placebo (Placebo Comparator): Placebo comparator
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Paliperidone — Paliperidone medication taken daily ranging from 3-9mg/day depending on tolerability and efficacy.
  Other Names: Invega
  Arms: Paliperidone
Drug: Placebo — Pill placebo taken daily ranging from 3-9mg/day depending on tolerability and efficacy.
  Arms: Pill placebo

SUMMARY:
Obsessive-compulsive disorder (OCD) is a common, chronic, and oftentimes disabling disorder. The only established treatments for OCD are a specific form of Cognitive Behavioral Therapy (CBT) and the Serotonin Reuptake Inhibitor medications (SRIs). Few patients with OCD experience complete symptom resolution with either modality and even after two consecutive SRI trials, as many as 30%-40% of patients fail to derive a satisfactory response. Pharmacological options for these SRI-resistant cases include switching to a different antidepressant, increasing the dose of SRI, or augmentation with another agent.

Previous studies showed that approximately 33-50% of OCD patients who have not had an adequate response to SRI medication had a positive response when an atypical antipsychotic medication was added. However, the problematic acute and long-term side effects of these medications are of concern and, at times, limit their use. Paliperidone has a number of advantages over these medications including fewer drug interactions and better tolerability. Thus, this study is designed to determine whether paliperidone augmentation of an existing medication is effective relative to taking a placebo and your existing medication.

DETAILED DESCRIPTION:
Obsessive-compulsive disorder (OCD) is a common, chronic, and oftentimes disabling disorder. The only established first-line treatments for OCD are a specific form of Cognitive Behavioral Therapy (CBT) and the Serotonin Reuptake Inhibitors (SRIs). Few patients with OCD experience complete symptom resolution with either modality. Even after two consecutive adequate SRI trials, as many as 30%-40% of patients fail to derive a satisfactory response. Pharmacological options for these SRI-resistant cases include switching to a different antidepressant, increasing the dose of SRI, or augmentation with another agent.

Among the pharmacological augmentation strategies, adjunctive antipsychotic medications enjoy the most empirical support as well as wide-scale use in clinical practice. Utilizing IMS Health's National Disease and Therapeutic Index (NDTI) for 12 months ending in November 2004, 4.2% of antipsychotic medication use is for anxiety and 1.3% specifically for OCD. Conversely, for OCD patients, antipsychotic medications account for 8.6% of drug use (IMS Health NDTI MAT, 2004). Among pediatric patients, prescriptions of antipsychotics increased from 8.6 out of 1,000 U.S. children in 1995-1996 to 39.4 out of 1,000 children in 2001-2002 (Cooper et al., 2006). Similarly, Medco, a private insurance company, noted that the rate of children 19 years and under covered by private insurance with at least one atypical prescription jumped 80% from 2001 to 2005 - from 3.6 per 1,000 to 6.5 per 1,000 (USA Today, extracted 5/2/2006). These rates parallel our own research, in which approximately 35% of adult patients on psychotropics were taking an antipsychotic in addition to their SRI. Thus, clearly there is a large sample of OCD patients that are being prescribed atypical antipsychotics to augment other treatments.

Previous studies showed that approximately 33-50% of OCD patients who have not had an adequate response to SRI medication had a positive response when an atypical antipsychotic medication was added (Bloch et al., 2006). Risperidone has been the most studied agent and has the most consistently positive findings (e.g., McDougle et al., 2000). However, the problematic acute and long-term side effects of risperidone (and other atypicals) are of concern and, at times, limit their use. Paliperidone, a metabolite of risperidone that utilizes OROS osmotic drug-release technology, has a number of advantages over risperidone including a lack of drug x drug interactions and a predictable pharmacokinetic profile that is associated with better tolerability. Thus, paliperidone has the potential to be a safer alternative for augmentation in OCD patients pending supporting efficacy data. Given the need to examine the efficacy of paliperidone, this protocol is designed to determine whether paliperidone augmentation of an SRI is effective relative to a placebo-control, and safe/tolerable in patients with OCD who have not adequately responded to past adequate SRI treatment.

ELIGIBILITY:
Inclusion Criteria:

1. Meets DSM-IV-TR criteria for a principal current diagnosis of OCD which is confirmed by both clinical evaluation and by structured interviews. OCD subjects with other comorbidities will be included provided OCD is judged to be the chief complaint.
2. Subjects must continue to experience clinically significant symptoms of OCD (Y-BOCS score ≥19 and a rating of "moderate" or greater on the Clinical Global Impressions (CGI) scale) despite at least two adequate SRI monotherapy trials. One unsatisfactory trial can include the SRI currently being taken by the patient provided that the duration of treatment is 12 weeks or more and that the dose has been adequate. Subjects must be taking a clinically effective dose of a SRI (i.e., clomipramine, citalopram, escitalopram, fluoxetine, fluvoxamine, paroxetine and sertraline) for at least 12 weeks. Subjects must be on their current dose for at least 12 weeks and must maintain their current dose throughout the study.
3. Between the ages of 18-70 years of age.
4. Only subjects with OC symptoms of at least one-year duration will be included.
5. Eligible subjects must be in good physical health. Screening procedures will include detailed medical history, complete physical and neurological exams, routine blood studies (CBC, liver function tests, electrolytes), ECG, urine toxicology screen, and serum pregnancy test in women of child-bearing potential.

Exclusion Criteria:

1. Primary depression, schizophrenia or other psychotic disorders.
2. Active bipolar disorder.
3. Non-responder in the past to atypical antipsychotic augmentation. This criterion was chosen to prevent recruiting a sample of chronically refractory OCD cases that would otherwise be suited for more extreme interventions such as deep brain stimulation.
4. Non-responder in the past to an adequate trial (> 20 hours) of cognitive-behavioral therapy that will be assessed by records review.
5. Current clinically significant suicidality or individuals who have engaged in suicidal behaviors within 6 months will be excluded and referred for appropriate clinical intervention.
6. Alcohol or other significant substance abuse within the last 6 months.
7. History of neurosurgery, encephalitis or significant head trauma or a significant medical condition such as heart, liver, or renal disease.
8. Nursing mothers or women of childbearing potential who do not use adequate contraception will be excluded.
9. Subjects at an increased risk for seizures will also be excluded from this study (e.g., subjects with a history of seizures [other than childhood febrile seizures], subjects taking concomitant medications known to lower the seizure threshold).
10. Estimated IQ < 80, mental retardation, dementia, brain damage, or other cognitive impairment that would interfere with the capacity to participate in the study and complete measures. If needed, the WASI will be used to assess this at screening.
11. Concurrent use of benzodiazepines, other than for treatment of insomnia, will be prohibited during the trial. No other psychotropic medications will be permitted.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2007-10; Primary Completion 2013-09 (Actual); Study Completion 2013-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Eric A Storch, Ph.D., Principal Investigator — University of South Florida
Locations (2):
- United States (2):
  - University of South Florida, St. Petersburg, Florida
  - University Hospital Outpatient Center, Psychiatry, Indianapolis, Indiana

REFERENCES:
- [Derived] Storch EA, Goddard AW, Grant JE, De Nadai AS, Goodman WK, Mutch PJ, Medlock C, Odlaug B, McDougle CJ, Murphy TK. Double-blind, placebo-controlled, pilot trial of paliperidone augmentation in serotonin reuptake inhibitor-resistant obsessive-compulsive disorder. J Clin Psychiatry. 2013 Jun;74(6):e527-32. doi: 10.4088/JCP.12m08278. PMID 23842022

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Thirty-four adults with a principal diagnosis of OCD were recruited between May 2008 and March 2012.
Groups:
- Paliperidone: Recieves study medication
  Paliperidone : Paliperidone medication taken daily ranging from 3-9mg/day depending on tolerability and efficacy.
- Placebo: Placebo comparator
  Paliperidone : Paliperidone medication taken daily ranging from 3-9mg/day depending on tolerability and efficacy.
Period: Overall Study
Arm/Group | Paliperidone | Placebo
Started | 17 | 17
Completed | 11 | 11
Not Completed | 6 | 6
Not completed — Adverse Event | 6 | 0
Not completed — Lost to Follow-up | 0 | 3
Not completed — Lack of Efficacy | 0 | 2
Not completed — Undisclosed reasons within the first wee | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Paliperidone | Placebo | Total
Number analyzed (Participants) | 17 | 17 | 34
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 17 | 16 | 33
  >=65 years | 0 | 1 | 1
Age, Continuous [Mean (Standard Deviation); unit: years] | 42.59 (9.99) | 45.7 (12.27) | 43.7 (11.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 9 | 10 | 19
  Male | 8 | 7 | 15
Region of Enrollment [Number; unit: participants]
  United States | 17 | 17 | 34

OUTCOME MEASURES:

1. Primary Outcome: Yale Brown Obsessive Compulsive Scale
Description: This measure assesses obsessive-compulsive symptom severity across 10 items that are completed during an interview format with the person with OCD. These 10 items are summed to derive a total score, which ranges from 0-40 [Scale range: 0 (Minimum) - 40 (Maximum)] with higher scores corresponding to more severe obsessive-compulsive symptoms.
Time Frame: End of study (8 weeks)
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Paliperidone | Placebo
Number analyzed (Participants) | 17 | 17
Scores on a scale | 19.14 (11.13) | 21.24 (8.16)
Statistical Analysis 1: Comparison: Paliperidone vs Placebo; To evaluate between-group continuous outcomes of the pilot controlled trial, ANCOVAs were performed, where 8-week outcome scores were predicted by treatment condition while covarying for baseline scores; Test type: Superiority or Other; p < 0.05, ANCOVA

2. Secondary Outcome: Clinical Global Impressions - Severity of Obsessive-Compulsive Symptoms
Description: This assessment measures the overall severity of obsessive-compulsive symptoms. It consists of a single item that is completed by a clinician with scores ranging from 0-6 with higher scores corresponding with more severe obsessive-compulsive symptoms. Thus, higher scores represent a worse outcome.
Time Frame: post-treatment
Population: Includes those subjects who were randomized to their respective condition.
Measure: Mean (Standard Deviation); unit: Scores on a scale
Arm/Group | Paliperidone | Placebo
Number analyzed (Participants) | 17 | 17
Scores on a scale | 4.09 (1.66) | 4.21 (1.29)
Statistical Analysis 1: Comparison: Paliperidone vs Placebo; [analysis description as in outcome 1, analysis 1]; Test type: Superiority or Other; p < 0.05, ANCOVA

ADVERSE EVENTS:
Time Frame: 8 weeks
Arm/Group | Paliperidone | Placebo
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/17
Other Adverse Events (participants affected / at risk) | 15/17 | 12/17
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Paliperidone (N=17) | Placebo (N=17)
Headache (Nervous system disorders) | 4 | 6
Dizziness (Nervous system disorders) | 3 | 4
Lightheadness (Nervous system disorders) | 3 | 3
blurred vision (Eye disorders) | 3 | 1
Muscle Stiffness (Nervous system disorders) | 4 | 0
Somnolence (General disorders) | 7 | 8
Insomnia (General disorders) | 5 | 5
Agitation (General disorders) | 4 | 2
Shakiness (Nervous system disorders) | 1 | 1
Anxiety (Psychiatric disorders) | 1 | 1
dry mouth (Gastrointestinal disorders) | 4 | 3
Nausea (Gastrointestinal disorders) | 0 | 3
Constipation (Gastrointestinal disorders) | 5 | 1
Increased need to urinate (Renal and urinary disorders) | 4 | 1
Ear Ringing (Ear and labyrinth disorders) | 2 | 2
Diarrhea (Gastrointestinal disorders) | 1 | 2
Galactorrhea (Reproductive system and breast disorders) | 2 | 0
Increased Appetite (Gastrointestinal disorders) | 5 | 3
Decreased Appetite (Gastrointestinal disorders) | 1 | 1

LIMITATIONS AND CAVEATS:
Modest sample and analyses were potentially underpowered to detect between-group differences on OCD measures.

It was not possible to determine response from participants' current medication.

Little racial/ethnic and socioeconomic variability

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No